CLINICAL TRIAL: NCT06031298
Title: Influence of Various Healing Intervals on Alveolar Ridge Preservation Using Demineralized Dentin Graft: A Randomized Clinical Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-REC 1254
Record Dates: First submitted 2023-09-02; First posted 2023-09-11 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Dentin Graft, Alveolar Ridge Preservation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alveolar ridge preservation using demineralized dentin graft at 12 weeks. (Experimental)
  Interventions: Biological: Dentin Graft
- Alveolar ridge preservation using demineralized dentin graft at 18 weeks (Active Comparator)
  Interventions: Biological: Dentin Graft
- Alveolar ridge preservation using demineralized dentin graft at 24 weeks (Active Comparator)
  Interventions: Biological: Dentin Graft

INTERVENTIONS:
Biological: Dentin Graft — Dentin graft is a grafting technique of autogenous origin that uses the teeth extracted from the patient for the graft material preparation.

SUMMARY:
Statement of the problem:

The alveolar ridge undergoes various remodeling processes following tooth extraction, but the ridge resorption continues over time, resulting in hard and soft tissue loss which complicates prosthodontic rehabilitation whether by dental implants or tooth supported prosthesis.

Aim of the study:

The aim of the study is to assess the influence of the different time intervals on the healing of the demineralized dentin graft in alveolar ridge preservation (ARP) procedures.

Materials and methods:

30 patients with hopeless teeth requiring extraction in maxillary non molar areas and requiring replacement with dental implants, will be enrolled and recruited from the outpatient clinic, faculty of dentistry, ain shams university according to the inclusion criteria. They will be randomly allocated into three equal groups. Group A (n=10) alveolar ridge preservation will be done with demineralized dentin graft and re-entry at 12 weeks, group B (n=10) alveolar ridge preservation will be done with demineralized dentin graft and re-entry at 18 weeks and group C (n=10) alveolar ridge preservation will be done with demineralized dentin graft and re-entry at 24 weeks. Radiographic assessment will be done using CBCT to the arch of interest and another cone beam will be done prior to the implant placement at 11, 17 and 23 weeks based on the study group and a volumetric assessment will be done with digital subtraction. At the respective times core biopsy will be taken for the histological assessment, and the implant placement will be done with the implant primary stability recorded using Ostell. Postoperative medication will be prescribed to the patient and postoperative instructions will be explained in detail. Follow-up will be performed. Data collected will be tabulated and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Systemically free patients (American Society of Anesthesiologists I; ASA I)
* Age range 20 - 50.
* Non-molar maxillary teeth indicated for extraction.
* Patients with extraction sockets having intact bony walls, or no more than one bony wall dehiscence not extending more than 50% of the total bone height

Exclusion Criteria:

* Teeth to be extracted or adjacent teeth associated with acute infections.
* Smokers.
* Patients with other conditions that may affect the treatment [uncontrolled diabetes mellitus (HbA1c >7.0), liver or kidney failure, any active oral or systemic acute infections, currently receiving chemo-or radiotherapy or a history of radiotherapy in the head and neck area, severe hematologic disorders].
* Pregnant and lactating females.
* Patients with history of lack of compliance to dental visits and unwillingness or inability to sign the informed consent.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic Assessment | Baseline, 12, 18 & 24 months
  Radiographic dimensional changes of the alveolar ridge following ARP using CBCT

SECONDARY OUTCOMES:
Implant primary stability | Time of implant placement at each group
  Implant primary stability using Ostell device
Histological Assessment | Core biopsy obtained at 12, 18 and 24 weeks for the different groups.
  Histomorphometric analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided